CLINICAL TRIAL: NCT05552963
Title: A Prospective, Multicenter, Single Arm With Performance Goal Study to Evaluate Safety and Effectiveness of Multi-electrode Circular IRE Catheter and Multi-Channel IRE Generator in Paroxysmal AF
Brief Title: A Study of Multi-electrode Circular Irreversible Electroporation (IRE) Catheter and Multi-Channel IRE Generator in Paroxysmal Atrial Fibrillation (AF)
Acronym: AFIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BWI202107; BWI202107 (Other: Biosense Webster, Inc.)
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Refractory Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electroporation; Radionuclide Generators

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Irreversible Electroporation (IRE) System (Experimental): Participants with symptomatic drug refractory paroxysmal atrial fibrillation (PAF) and indicated for catheter ablation will be treated with the IRE system which includes multi-electrode circular IRE catheter and the multi-channel IRE generator.
  Interventions: Device: Multi-Channel Irreversible Electroporation (IRE) Generator; Device: Multi-Channel Circular IRE Catheter

INTERVENTIONS:
Device: Multi-Channel Irreversible Electroporation (IRE) Generator — The multi-channel IRE Generator is intended for use during cardiac Pulsed Field Ablation (PFA) therapy. This device is used in conjunction with a compatible ablation catheter to create a closed electrical circuit capable of delivering pulsed electrical field energy.
  Other Names: D-1417-01-I
Device: Multi-Channel Circular IRE Catheter — The multi-channel circular IRE Catheter is indicated for use in catheter-based cardiac electrophysiological mapping (stimulating and recording) and when used with an IRE Generator, for cardiac ablation.
  Other Names: D-1412-01-SI

SUMMARY:
The purpose of this study is to evaluate the long term off-Antiarrhythmic Drug (AAD) effectiveness of Biosense Webster, Inc. Irreversible Electroporation (BWI IRE) system in treatment of participants with symptomatic drug refractory paroxysmal atrial fibrillation (PAF).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with symptomatic paroxysmal atrial fibrillation (PAF) (Physician's note indicating recurrent self-terminating atrial fibrillation [AF]). At least one electrocardiographically documented AF episode within twelve (12) months prior to enrollment. Electrocardiographic documentation may include, but is not limited to, electrocardiogram (ECG), Holter monitor, or telemetry strip
* Failed at least one Class I or Class III antiarrhythmic drug (AAD) as evidenced by recurrent symptomatic AF, contraindicated or intolerable to both Class I and Class III AAD
* Able and willing to comply with all pre-procedure, post-procedure, and follow-up testing and visit requirements
* Willing and capable of providing consent

Exclusion Criteria:

* AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause (Example, untreated documented obstructive sleep apnea and acute alcohol toxicity)
* Previous left atrium (LA) ablation or surgery
* Participants known to require ablation outside the pulmonary vein (PV) region (atrioventricular reentrant tachycardia, atrioventricular nodal reentry tachycardia, atrial tachycardia, atrial flutter of unknown origin, ventricular tachycardia and Wolff-Parkinson-White)
* Previously diagnosed with persistent AF (greater than [>] 7 days in duration)
* Severe dilatation of the LA (documented LAD >50 millimeters [mm] antero-posterior diameter by transthoracic echocardiography (TTE) within 6 month prior to enrollment)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jianzeng Dong, Study Chair — The First Affiliated Hospital of Zhengzhou University; Shaowen Liu, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine; Hailong Tao, Principal Investigator — The First Affiliated Hospital of Zhengzhou University; Hua Fu, Principal Investigator — West China Hospital; Yumei Xue, Principal Investigator — Guangdong Provincial People's Hospital; Heng Cai, Principal Investigator — Tianjin Medical University General Hospital; Lianjun Gao, Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (6):
- China (6):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The first affiliated hospital of Zhengzhou University, Zhengzhou, Henan
  - The first affiliated hospital of Dalian Medical University, Dalian, Liaoning
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Irreversible Electroporation (IRE) System: Participants with symptomatic drug refractory paroxysmal atrial fibrillation (PAF) and indicated for catheter ablation were treated with the IRE system which included multi-electrode circular IRE catheter and the multi-channel IRE generator.
Period: Overall Study
Arm/Group | Irreversible Electroporation (IRE) System
Started | 142
Roll-in Participants | 19
Non-roll-in Participants | 123
Completed the Index Ablation Procedure | 142
Completed | 140
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Study catheter was inserted, but PF energy was not delivered due to ECG interference | 1

BASELINE CHARACTERISTICS:
Arm/Group | Irreversible Electroporation (IRE) System
Number analyzed (Participants) | 142
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.9 (12.04)
Age, Customized [Count of Participants; unit: Participants]
  <45 years | 26
  Between 45 to <65 years | 67
  >=65 years | 49
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 81
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Long-term Effectiveness
Description: Long-term effectiveness was defined as freedom from documented asymptomatic and symptomatic atrial fibrillation (AF), atrial tachycardia (AT), or atrial flutter (AFL; of unknown origin) episodes based on electrocardiographic data (greater than equal to [>=] 30 seconds on arrhythmia monitoring device) through the effectiveness evaluation period (Day 91 through Day 365 post index procedure) and freedom from the following failure modes : freedom from acute procedural failure, freedom from non-study catheter failure, freedom from repeat ablation failure, freedom from direct Current (DC) cardioversion failure, freedom from recurrence (captured on 12-lead electrocardiogram [ECG]) failure, and freedom from anti-arrhythmic drug failure. AFL of unknown origin was defined as all AFL except those Cavo-Tricuspid Isthmus (CTI) dependent AFL as confirmed by accepted electrophysiology (EP) maneuvers (for example, entrainment or activation mapping) in an EP study.
Time Frame: From Day 91 up to Day 365 post-procedure on Day 0
Population: Full analysis set (FAS) included all enrolled non-roll-in participants who were ablated with investigational devices. Here, 'N' (overall number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Irreversible Electroporation (IRE) System
Number analyzed (Participants) | 122
Percentage of participants | 74.6 [66.86 to 82.32]

2. Secondary Outcome: Percentage of Participants Experiencing Primary Adverse Event (PAE)
Description: Percentage of participants experiencing PAE were reported. An AE is any untoward medical occurrence in a participant whether or not related to the investigational medical device. Primary AEs within seven days of the ablation procedure which used investigational devices per protocol, including the initial and repeat procedures were reported. PAEs included cardiac tamponade, perforation, myocardial infarction, stroke/cerebrovascular accident, thromboembolism, transient ischaemic attack, phrenic nerve injury/diaphragmatic paralysis, heart block, pulmonary vein stenosis, pulmonary oedema (respiratory insufficiency), vagal nerve injury/gastroparesis, pericarditis, major vascular access complication/bleeding, and atrio-esophageal fistula .
Time Frame: Within 7 days post-procedure on Day 0
Population: Safety analysis set included all the enrolled participants (including both non roll-in and roll-in participants) who had the investigational devices inserted or treated.
Measure: Number; unit: Percentage of participants
Arm/Group | Irreversible Electroporation (IRE) System
Number analyzed (Participants) | 142
Percentage of participants | 2.1

3. Secondary Outcome: Percentage of Participants Experiencing Serious Adverse Event (SAE) Within 7 Days, 8-30 Days and >30 Days of Initial Ablation Procedure
Description: Percentage of participants with SAEs within 7 days (early-onset), 8-30 days (peri-procedural) and >30 days (late onset) of initial ablation procedure were reported. A SAE was any adverse event (AE) that resulted in a death or a serious deterioration in the health of the participant during the clinical trial, including a life-threatening illness or injury, a permanent impairment of a body structure or a body function, in-patient hospitalization or prolongation of existing hospitalization, medical or surgical intervention to prevent permanent impairment of a body structure or a body function; or resulted in fetal distress, foetal death or congenital abnormality, congenital anomaly, etc.
Time Frame: From day of procedure (Day 0) up to 12 months
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Irreversible Electroporation (IRE) System
Number analyzed (Participants) | 142
Percentage of participants
  Within 7 days (early-onset) of index ablation procedure | 2.8
  Within 8-30 days (peri-procedural) | 0.7
  >30 days (late onset) | 6.3

4. Secondary Outcome: Percentage of Participants With Acute Procedural Success
Description: Percentage of participants with acute procedural success were reported. Acute procedural success was defined as confirmation of entrance block in all clinically relevant targeted pulmonary veins (PVs) after adenosine/ isoproterenol challenge. Touching up with focal catheter was considered as acute procedural failure.
Time Frame: On the day of procedure (Day 0)
Population: Full analysis set (FAS) included all enrolled non-roll-in participants who were ablated with investigational devices.
Measure: Number; unit: Percentage of participants
Arm/Group | Irreversible Electroporation (IRE) System
Number analyzed (Participants) | 123
Percentage of participants | 100

5. Secondary Outcome: Percentage of Participants With Acute Reconnection
Description: Percentage of participants with acute reconnection were reported. Acute reconnection was identified by adenosine/isoproterenol challenge among all clinically relevant targeted PVs and by participant.
Time Frame: On the day of procedure (Day 0)
Population: Full analysis set (FAS) included all enrolled non-roll-in participants who were ablated with investigational devices.
Measure: Number; unit: Percentage of participants
Arm/Group | Irreversible Electroporation (IRE) System
Number analyzed (Participants) | 123
Percentage of participants | 10.6

6. Secondary Outcome: Percentage of Pulmonary Veins (PVs) With Acute Reconnection
Description: Percentage of PVs with acute reconnection were reported. Acute reconnection was identified by adenosine/isoproterenol challenge among all clinically relevant targeted PVs and by participant.
Time Frame: On the day of procedure (Day 0)
Population: Full analysis set (FAS) included all enrolled non-roll-in participants who were ablated with investigational devices.
Measure: Number; unit: Percentage of pulmonary veins
Units Other Than Participants: Pulmonary veins
Arm/Group | Irreversible Electroporation (IRE) System
Number analyzed (Participants) | 123
Number analyzed (Pulmonary veins) | 490
Percentage of pulmonary veins | 4.7

7. Secondary Outcome: Percentage of Participants With Pulmonary Vein (PV) Ablation
Description: Percentage of participants with PV ablation by a non-study catheter (touch-up) among all clinically relevant targeted participants were reported.
Time Frame: On day of procedure (Day 0)
Population: Full analysis set (FAS) included all enrolled non-roll-in participants who were ablated with investigational devices.
Measure: Number; unit: Percentage of participants
Arm/Group | Irreversible Electroporation (IRE) System
Number analyzed (Participants) | 123
Percentage of participants | 0 [8.52 to 75.51]

8. Secondary Outcome: Percentage of Participants With Repeated Ablation
Description: Percentage of participants with repeated ablation within the 12 months follow up period, including timing (blanking period or after blanking) were reported. Repeat procedures for AF/AT/AFL of unknown origin plus recurrences during the blanking period (90 days post index procedure) were conducted with the investigational device for ablating PV reconnections. Repeat procedures performed after the blanking period were managed per investigator discretion using a commercially available ablation catheter and generator.
Time Frame: From the day of procedure (Day 0) up to 12 months
Population: Full analysis set (FAS) included all enrolled non-roll-in participants who were ablated with investigational devices.
Measure: Number; unit: Percentage of participants
Arm/Group | Irreversible Electroporation (IRE) System
Number analyzed (Participants) | 123
Percentage of participants | 6.5

ADVERSE EVENTS:
Time Frame: From the time of informed consent signing through 12 months post-procedure (on Day 0)
Description: Safety analysis set included all the enrolled participants (including both non roll-in participants and roll-in participants) who had the investigational devices inserted or treated.
Arm/Group | Irreversible Electroporation (IRE) System
All-Cause Mortality (participants affected / at risk) | 0/142
Serious Adverse Events (participants affected / at risk) | 16/142
Other Adverse Events (participants affected / at risk) | 13/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Irreversible Electroporation (IRE) System (N=142)
Upper respiratory tract infection (Infections and infestations) | 2
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Generalised anxiety disorder (Psychiatric disorders) | 1
Obsessive-compulsive disorder (Psychiatric disorders) | 1
Arteriovenous fistula (Vascular disorders) | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1
Puncture site haematoma (General disorders) | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Vitreous haemorrhage (Eye disorders) | 1
Cataract nuclear (Eye disorders) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1
Device dislocation (Product Issues) | 1
Vertigo (Ear and labyrinth disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Irreversible Electroporation (IRE) System (N=142)
Upper respiratory tract infection (Infections and infestations) | 11
COVID-19 (Infections and infestations) | 5
Nausea (Gastrointestinal disorders) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Supraventricular tachycardia (Cardiac disorders) | 5
Dysuria (Renal and urinary disorders) | 9
Haematuria (Renal and urinary disorders) | 5
Insomnia (Psychiatric disorders) | 5
Blood pressure increased (Investigations) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/63/NCT05552963/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT05552963/SAP_001.pdf